CLINICAL TRIAL: NCT00849901
Title: A Double-Blind, Efficacy and Safety Study of Duloxetine Versus Placebo in the Treatment of Children and Adolescents With Major Depressive Disorder
Brief Title: A Study in the Treatment of Children and Adolescents With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6223; F1J-MC-HMCK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fluoxetine (Active Comparator)
  Interventions: Drug: fluoxetine
- Duloxetine (Experimental)
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — 30-120 mg, PO, QD, for up to 38 weeks
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — Capsules identical in appearance, color, taste and smell to study drug, orally (PO), once daily (QD). Dose: placebo, 6 capsules, QD for 10 weeks
  Arms: Placebo
Drug: fluoxetine — 10-40 milligram (mg), PO, QD, for up to 38 weeks
  Other Names: LY110140; Prozac
  Arms: Fluoxetine

SUMMARY:
The purpose of this study is to assess whether duloxetine is superior to placebo in the treatment of children and adolescents with major depressive disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, diagnosed with major depressive disorder (MDD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and supported by the Mini International Neuropsychiatric Interview for children and adolescents (MINI-KID).
* Diagnosis of moderate or greater severity of MDD as determined by Children's Depression Rating Scale - Revised (CDRS-R) with a total score greater than or equal to 40 at screen, and randomization and a Clinical Global Impression of Severity (CGI-Severity) rating of greater than or equal to 4 at screen, and randomization.
* Female patients must test negative for pregnancy during screening.
* Judged to be reliable by the investigator to keep all appointments for clinical visits, tests, and procedures required by the protocol.
* Has a degree of understanding such that they can communicate intelligently with the investigator and study coordinator.
* Capable of swallowing study drug whole. It is anticipated the patients will need to swallow up to 6 capsules per day.
* Patients must have venous access sufficient to allow blood sampling and are compliant with blood draws as per the protocol.

Exclusion Criteria:

* Children of site personnel directly affiliated with this study and/or their immediate families.
* Children of Lilly employees or employees of the designated clinical research organization (CRO) assisting with the conduct of the study.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, or pervasive development disorder, as judged by the investigator.
* Have a history of DSM-IV-TR-defined substance abuse or dependence within the past year, excluding caffeine and nicotine.
* Have a current primary DSM-IV-TR Axis I disorder other than MDD or a current secondary DSM-IV-TR Axis I disorder that requires any pharmacologic treatment
* Have 1 or more first-degree relatives with diagnosed bipolar I disorder.
* Have a significant suicide attempt within 1 year of screening or are currently at risk of suicide in the opinion of the investigator.
* Have a weight less than 20 kilogram (kg) at screening.
* Have a lack of response to 2 or more adequate treatment trials of antidepressants at a clinically appropriate dose for a minimum of 4 weeks for the same MDD episode.
* Have initiated, stopped, or changed the type or intensity of psychotherapy within 6 weeks prior to screening.
* Have a history of seizure disorder (other than febrile seizures).
* Have a history of electroconvulsive therapy within 1 year of screening.
* Have had treatment with a monoamine oxidase inhibitor (MAOI) within 14 days or fluoxetine within 30 days of randomization; or the potential need to use an MAOI during the study or within 5 weeks of discontinuation of study drug.
* Have previously enrolled, completed, or withdrawn from this study or any other study investigating duloxetine or fluoxetine.
* Have a positive urine drug screen for any substances of abuse or excluded medication.
* Are taking any excluded medications that cannot be discontinued by screening.
* Have known hypersensitivity to duloxetine, fluoxetine, or their inactive ingredients; or have frequent or severe allergic reactions to multiple medications.
* Have uncontrolled narrow-angle glaucoma.
* Have acute liver injury or severe cirrhosis.
* Have a serious or unstable medical illness, psychological condition, or clinically significant laboratory or electrocardiogram (ECG) result that, in the opinion of the investigator, would compromise participation in the study or be likely to lead to hospitalization.
* Have abnormal thyroid-stimulating hormone concentration.
* Have initiated or discontinued hormone therapy within the previous 3 months.
* Female patients who are either pregnant, nursing or have recently given birth.
* Need to use thioridazine during the study or within 5 weeks after discontinuation of study drug or need to use pimozide during the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 337 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (59):
- United States (24):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Costa Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Altamonte Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smyrna, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coeur d'Alene, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Charles, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willingboro, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bartlett, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orem, Utah
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Élancourt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouffach
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Russia (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kazan'
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolensk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomsk
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Martin
- South Africa (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Centurion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vereeniging
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Cape
- Ukraine (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luhansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ternopil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uzhhorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

REFERENCES:
- [Derived] Emslie GJ, Wells TG, Prakash A, Zhang Q, Pangallo BA, Bangs ME, March JS. Acute and longer-term safety results from a pooled analysis of duloxetine studies for the treatment of children and adolescents with major depressive disorder. J Child Adolesc Psychopharmacol. 2015 May;25(4):293-305. doi: 10.1089/cap.2014.0076. PMID 25978741
- [Derived] Atkinson SD, Prakash A, Zhang Q, Pangallo BA, Bangs ME, Emslie GJ, March JS. A double-blind efficacy and safety study of duloxetine flexible dosing in children and adolescents with major depressive disorder. J Child Adolesc Psychopharmacol. 2014 May;24(4):180-9. doi: 10.1089/cap.2013.0146. Epub 2014 May 9. PMID 24813026
- [Derived] Bliznak L, Berg R, Hage A, Dittmann RW. High rate of non-eligibility: methodological factors impacting on recruitment for a multicentre, double-blind study of paediatric patients with major depressive disorder. Pharmacopsychiatry. 2013 Jan;46(1):23-8. doi: 10.1055/s-0032-1314806. Epub 2012 Jun 14. PMID 22699956

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a 10-week acute treatment phase, and a 6-month extension phase.
Groups:
- Duloxetine/Duloxetine: Received duloxetine 60, 90, and/or 120 milligram (mg) orally (PO), once daily (QD) during both acute treatment phase and extension phase
- Fluoxetine/Fluoxetine: Received fluoxetine 20 and/or 40 mg PO, QD during both acute treatment phase and extension phase
- Placebo/Duloxetine: Received placebo PO, QD during acute treatment phase, and duloxetine 60, 90, and/or 120 mg PO, QD during extension phase
Period: Acute Treatment Phase
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Started | 117 | 117 | 103
Completed | 87 (4 didn't enter extension phase.) | 91 | 87 (1 didn't enter extension phase.)
Not Completed | 30 | 26 | 16
Not completed — Adverse Event | 9 | 1 | 3
Not completed — Lost to Follow-up | 2 | 4 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 10 | 4
Not completed — Parent or Caregiver Decision | 11 | 5 | 4
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 2
Period: Extension Phase
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Started | 83 | 91 | 86
Completed | 56 | 65 | 69
Not Completed | 27 | 26 | 17
Not completed — Adverse Event | 2 | 8 | 4
Not completed — Lost to Follow-up | 3 | 0 | 1
Not completed — Protocol Violation | 2 | 2 | 4
Not completed — Withdrawal by Subject | 7 | 6 | 3
Not completed — Parent or Caregiver Decision | 10 | 4 | 4
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Lack of Efficacy | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine | Total
Number analyzed (Participants) | 117 | 117 | 103 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.14 (3.043) | 13.08 (3.272) | 13.28 (3.055) | 13.16 (3.120)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 51 | 176
  Male | 53 | 56 | 52 | 161
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 2 | 0 | 2
  Black or African American | 17 | 9 | 13 | 39
  White | 90 | 93 | 79 | 262
  Multiracial | 4 | 7 | 5 | 16
  Not Provided | 5 | 5 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 50 | 45 | 45 | 140
  Finland | 1 | 4 | 0 | 5
  France | 3 | 2 | 3 | 8
  Germany | 1 | 1 | 2 | 4
  Slovakia | 2 | 3 | 1 | 6
  Ukraine | 25 | 23 | 18 | 66
  Russian Federation | 13 | 15 | 12 | 40
  Estonia | 1 | 0 | 0 | 1
  South Africa | 21 | 24 | 22 | 67
Children's Depression Rating Scale-Revised (CDRS-R) Total Score [Mean (Standard Deviation); unit: units on a scale] — CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression.
  units on a scale | 59.2 (10.45) | 58.8 (10.56) | 60.2 (11.67) | 59.4 (10.85)
CDRS-R Subscale Scores [Mean (Standard Deviation); unit: units on a scale] — CDRS-R Subscale score include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21.
  units on a scale
    Mood | 16.3 (3.54) | 15.9 (3.85) | 16.1 (3.59) | 16.1 (3.66)
    Somatic | 19.8 (4.54) | 19.7 (4.21) | 20.0 (4.75) | 19.8 (4.48)
    Subjective | 10.1 (3.08) | 10.4 (3.24) | 10.4 (3.46) | 10.3 (3.25)
    Behavior | 13.0 (2.79) | 12.8 (2.87) | 13.5 (3.00) | 13.1 (2.89)
Clinical Global Impressions of Severity (CGI-Severity) score [Mean (Standard Deviation); unit: units on a scale] — CGI-Severity score evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 4.5 (0.62) | 4.5 (0.58) | 4.6 (0.65) | 4.5 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 10 Endpoint
Description: CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. Least Square (LS) means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: Received duloxetine 60, 90, and/or 120 mg orally (PO), once daily (QD) during acute treatment phase
- Fluoxetine: Received fluoxetine 20 and/or 40 mg PO, QD during acute treatment phase
- Placebo: Received placebo PO, QD during acute treatment phase
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 113 | 113 | 103
units on a scale | -24.3 (1.09) | -23.7 (1.06) | -24.3 (1.11)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis

2. Secondary Outcome: Change From Week 10 in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at Week 36 Endpoint
Description: CDRS-R Total score measure the presence and severity of depression in children. The scale consists of 17 items scored on a 1-to-5- or 1-to-7-point scale. A rating of 1 indicates normal functioning. Total scores range from 17 to 113. In general, scores below 20 indicate an absence of depression, scores of 20 to 30 indicate borderline depression, and scores of 40 to 60 indicate moderate depression. LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 81 | 91 | 85
units on a scale | -7.2 (0.86) | -9.9 (0.72) | -9.6 (0.86)

3. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Subscale Score at Week 10 Endpoint
Description: CDRS-R Subscale scores include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21. Higher score indicates greater severity of disease. LS means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 113 | 113 | 103
units on a scale
  Mood (N=113, 113, 103) | -7.0 (0.36) | -7.1 (0.35) | -7.0 (0.37)
  Somatic (N=113, 113, 103) | -7.7 (0.42) | -7.6 (0.41) | -7.7 (0.42)
  Subjective (N=113, 113, 103) | -4.0 (0.23) | -3.6 (0.22) | -4.0 (0.23)
  Behavior (N=113, 112, 103) | -5.6 (0.30) | -5.4 (0.30) | -5.7 (0.31)

4. Secondary Outcome: Change From Week 10 in Children's Depression Rating Scale-Revised (CDRS-R) Subscale Score at Week 36 Endpoint
Description: CDRS-R Subscale scores include Mood (Sum of items 8, 11, 14, 15), Somatic (Sum of items 4-7, 16, 17), Subjective (Sum of items 9, 10, 12, 13) and Behavior (Sum of items 1-3). Mood and Subjective subscale scores range from 4 to 28; Somatic subscale scores range from 6 to 36; Behavior subscale scores range from 3 to 21. Higher score indicates greater severity of disease. LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 81 | 91 | 85
units on a scale
  Mood | -1.9 (0.34) | -2.5 (0.24) | -2.9 (0.29)
  Somatic | -2.8 (0.35) | -3.6 (0.27) | -3.2 (0.33)
  Subjective | -0.3 (0.24) | -1.3 (0.13) | -1.2 (0.17)
  Behavior | -1.9 (0.23) | -2.8 (0.20) | -2.1 (0.36)

5. Secondary Outcome: Change From Baseline in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 10 Endpoint
Description: CGI-Severity evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS means are adjusted for baseline, pooled investigator, age category, visit, treatment, treatment*visit, age category*visit and baseline*visit.
Time Frame: Baseline, Week 10
Population: Participants with both a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 113 | 113 | 110
units on a scale | -1.9 (0.11) | -1.8 (0.10) | -1.9 (0.11)

6. Secondary Outcome: Change From Week 10 in Clinical Global Impressions of Severity (CGI-Severity) Scale at Week 36 Endpoint
Description: CGI-Severity evaluates the severity of illness at the time of assessment. The score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). LS means are adjusted for baseline, pooled investigator, age category, visit, age category*visit and baseline*visit.
Time Frame: Week 10, Week 36
Population: Participants with value during treatment phase and at least one post-Week 10 value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 81 | 91 | 85
units on a scale | -0.6 (0.12) | -1.0 (0.07) | -1.1 (0.10)

7. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior Baseline Through Week 10
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Treatment Emergent Suicidal Ideation is worsening or new occurrence of events during treatment compared to lead-in baseline (Week -1 - 0).
Time Frame: Baseline through Week 10
Population: Participants with at least one post-baseline C-SSRS suicidal ideation or suicidal behavior score and who are at risk for treatment emergent suicidal ideation or behavior.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 113 | 113 | 103
participants
  Suicidal Ideation | 16 | 16 | 15
  Suicidal Behavior | 0 | 1 | 0
  Treatment Emergent Suicidal Ideation | 8 | 9 | 7

8. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior Week 10 Through Week 36
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Treatment Emergent Suicidal Ideation is worsening or new occurrence of events during treatment compared to lead-in baseline (Week 7-10).
Time Frame: Week 10 through Week 36
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 81 | 91 | 85
participants
  Suicidal Ideation | 13 | 13 | 8
  Suicidal Behavior | 1 | 1 | 0
  Treatment Emergent Suicidal Ideation | 9 | 13 | 8

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hepatic Laboratory Results Any Time Baseline Through Week 10
Description: Total number of participants with any abnormal post-baseline value, based on all values at scheduled and unscheduled visits. Potentially clinically significant hepatic laboratory results at any time are defined as alanine transaminase (ALT) ≥3 x upper limit of normal (ULN), ALT ≥5 x ULN and ALT ≥10 x ULN, as well as ALT ≥3 x ULN and Total Bilirubin ≥2 x ULN.
Time Frame: Baseline through Week 10
Population: Participants with normal ALT value (ALT <1 x ULN) at last non-missing baseline visit and at least one non-missing post-baseline value.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 101 | 102 | 94
participants
  ALT≥3 x ULN | 0 | 0 | 0
  ALT≥5 x ULN | 0 | 0 | 0
  ALT≥10 x ULN | 0 | 0 | 0
  ALT≥3 x ULN and Total Bilirubin≥2 x ULN | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hepatic Laboratory Results Any Time Week 10 Through Week 36
Description: as for outcome 9
Time Frame: Week 10 through Week 36
Population: Participants with normal ALT value (ALT<1 x ULN) at last non-missing visit before Week 10 and at least one non-missing post-Week 10 value.
Measure: Number; unit: participants
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 77 | 83 | 82
participants
  ALT≥3 x ULN | 0 | 1 | 0
  ALT≥5 x ULN | 0 | 1 | 0
  ALT≥10 x ULN | 0 | 0 | 0
  ALT≥3 x ULN and Total Bilirubin≥2 x ULN | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Changes in Systolic Blood Pressure (BP), Diastolic BP, Pulse, and Weight Any Time Baseline Through Week 10
Description: PCS increase in systolic and diastolic BP was defined as increase of ≥5 millimeter mercury (mm Hg) from baseline (BL) high value to a value above the 95th percentile at post-BL; PCS increase of pulse was defined as >140 and increase of ≥15 from BL high value for age 7-11 and >120 and increase of ≥15 from BL high value for age 12-17; PCS decrease of pulse was defined as <60 and a decrease of ≥25 from BL low value for age 7-11 and <50 and a decrease of ≥15 from BL low value for age 12-17; PCS decrease of weight was defined as decrease of at least 3.5% from BL low value.
Time Frame: Baseline through Week 10
Population: Participants with normal baseline value and at least one post-baseline value, and who were at risk for the specific PCS criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Fluoxetine | Placebo
Number analyzed (Participants) | 117 | 117 | 103
percentage of participants
  Diastolic BP Increase (N=102, 106, 93) | 8.8 | 7.5 | 17.2
  Systolic BP Increase (N=100, 106, 90) | 7.0 | 5.7 | 6.7
  Pulse Decrease (N=111, 112, 102) | 0.9 | 0.9 | 1.0
  Pulse Increase (N=113, 114, 103) | 0 | 0 | 1.0
  Weight Decrease (N=113, 114, 103) | 12.4 | 11.4 | 4.9

12. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant (PCS) Changes in Systolic Blood Pressure (BP), Diastolic BP, Pulse, and Weight Any Time Week 10 Through Week 36
Description: PCS increase in systolic and diastolic BP was defined as increase of ≥ 5mm Hg from baseline (BL) high value to a value above the 95th percentile at post-BL; PCS increase of pulse was defined as >140 and increase of ≥15 from BL high value for age 7-11 and >120 and increase of ≥15 from BL high value for age 12-17; PCS decrease of pulse was defined as <60 and a decrease of ≥25 from BL low value for age 7-11 and <50 and a decrease of ≥15 from BL low value for age 12-17; PCS decrease of weight was defined as decrease of at least 3.5% from BL low value.
Time Frame: Week 10 through Week 36
Population: Participants with normal value at last non-missing visit before Week 10 and at least one non-missing post-Week 10 value, and who are at risk for the specific PCS criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine/Duloxetine | Fluoxetine/Fluoxetine | Placebo/Duloxetine
Number analyzed (Participants) | 83 | 91 | 86
percentage of participants
  Diastolic BP Increase (N=65, 76, 61) | 16.9 | 11.8 | 4.9
  Systolic BP Increase (N=64, 80, 69) | 12.5 | 12.5 | 10.1
  Pulse Decrease (N=78, 84, 82) | 0 | 0 | 0
  Pulse Increase (N=81, 91, 84) | 0 | 0 | 0
  Weight Decrease (N=81, 91, 85) | 6.2 | 3.3 | 9.4

ADVERSE EVENTS:
Groups:
- Duloxetine - Acute: Received duloxetine 60, 90, and/or 120 mg orally (PO), once daily (QD) during acute treatment phase
- Fluoxetine - Acute: Received fluoxetine 20 and/or 40 mg PO, QD during acute treatment phase
- Placebo - Acute: Received placebo PO, QD during acute treatment phase
- Duloxetine - Extension; Placebo/Duloxetine - Extension: Received duloxetine 60, 90, and/or 120 mg PO, QD during extension phase
- Fluoxetine - Extension: Received fluoxetine 20 and/or 40 mg PO, QD during extension phase. One participant had discontinued the acute phase due to an adverse event but was accidentally dispensed drug at the last visit of the acute phase, thus based on intent-to-treat principal, this participant was included in the extension phase analyses for adverse events (AEs) (resulting in one more participant being analyzed for AEs than started the extension phase in the Participant Flow section).
Arm/Group | Duloxetine - Acute | Fluoxetine - Acute | Placebo - Acute | Duloxetine - Extension | Fluoxetine - Extension | Placebo/Duloxetine - Extension
Serious Adverse Events (participants affected / at risk) | 3/117 | 2/117 | 1/103 | 1/83 | 4/92 | 4/86
Other Adverse Events (participants affected / at risk) | 70/117 | 72/117 | 68/103 | 53/83 | 56/92 | 60/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Acute (N=117) | Fluoxetine - Acute (N=117) | Placebo - Acute (N=103) | Duloxetine - Extension (N=83) | Fluoxetine - Extension (N=92) | Placebo/Duloxetine - Extension (N=86)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with disturbance of conduct (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Social phobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Acute (N=117) | Fluoxetine - Acute (N=117) | Placebo - Acute (N=103) | Duloxetine - Extension (N=83) | Fluoxetine - Extension (N=92) | Placebo/Duloxetine - Extension (N=86)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 5 (7) | 7 (8) | 1 (1) | 2 (2) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 20 (28) | 15 (17) | 11 (14) | 3 (6) | 7 (8) | 12 (17)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (7) | 3 (3) | 4 (5) | 5 (5) | 8 (9)
Fatigue (General disorders) | 8 (8) | 3 (5) | 5 (5) | 1 (1) | 3 (3) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 7 (7) | 3 (3) | 6 (8) | 5 (6) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 5 (5) | 9 (9) | 8 (12) | 9 (9)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 5 (6) | 5 (7) | 3 (3)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 3 (3) | 4 (5) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11) | 10 (10) | 7 (7) | 2 (3) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 10 (11) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 19 (23) | 18 (22) | 9 (10) | 9 (10) | 9 (10) | 10 (12)
Somnolence (Nervous system disorders) | 7 (7) | 6 (6) | 6 (6) | 2 (2) | 4 (5) | 3 (4)
Insomnia (Psychiatric disorders) | 6 (8) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days